CLINICAL TRIAL: NCT05826457
Title: North American Prodromal Synucleinopathy Consortium Stage 2
Acronym: NAPS2
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Mayo Clinic (Other); University of Minnesota (Other); University of California, Los Angeles (Other); McGill University (Other); Emory University (Other); Massachusetts General Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Stanford University (Other); National Institutes of Health (NIH) (NIH); Oregon Health and Science University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1234567; U19AG071754 (NIH)
Record Dates: First submitted 2023-02-08; First posted 2023-04-24 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: REM Sleep Behavior Disorder; Parkinson Disease; Lewy Body Dementia; Dementia With Lewy Bodies; Multiple System Atrophy; REM Sleep Parasomnias
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease; Lewy Body Disease; Multiple System Atrophy; REM Sleep Parasomnias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, buffy coat, paxgene, and cerebral spinal fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RBD group: Clinical observation involving annual visits to a study site for up to 5 years.
- control group: Clinical observation involving annual visits to a study site for up to 5 years.

SUMMARY:
This study will enroll participants with idiopathic REM sleep behavior disorder (RBD) and healthy controls for the purpose of preparing for a clinical trial of neuroprotective treatments against synucleinopathies.

DETAILED DESCRIPTION:
REM sleep behavior disorder (RBD) is a disorder where people act out their dreams. People with RBD often, but not always, develop Parkinson's Disease, dementia with Lewy bodies, multiple system atrophy, or other neurodegenerative diseases of the synucleinopathy type.

The North American Prodromal Synucleinopathy Consortium Stage 2 (NAPS2) was formed with the purpose of enrolling participants with RBD, in anticipation of a future clinical trial of a neuroprotective trreatment against synucleinopathies. The NAPS Consortium will collect standardized clinical assessments, biofluids, and neuroimaging data. The RBD group will also undergo two overnight sleep studies. Some of this data will be used to develop biomarkers for synucleinopathies in the prodromal (presymptomatic) stage as well as a trial-ready registry of participants.

RBD group procedures include a clinical assessment, questionnaires, blood draw, neuroimaging (MRI and DaTscan), polysomnogram (sleep study), and optional lumbar puncture.

Control group procedures include a clinical assessment, questionnaires, blood draw, neuroimaging (MRI), and lumbar puncture.

ELIGIBILITY:
Inclusion Criteria for RBD Group

1. Polysomnogram-confirmed RBD by ICSD-3 criteria
2. Capable of providing informed consent at time of study enrollment
3. Age > 18 years

Exclusion Criteria for RBD Group

1. Diagnosis of PD, dementia of any type, or MSA unless previous participant in NAPS1.
2. Narcolepsy-associated RBD
3. RBD secondary to any known cause except prodromal synucleinopathy.
4. Participation in a clinical trial, except by specific permission by the Executive Committee
5. In the opinion of the investigator, the individual has a clinically significant uncontrolled medical condition that would impede safe completion of the study protocol

Inclusion Criteria for Control Group

1. Ability to provide written consent
2. Age > 18 years
3. Must meet age, sex, and race matching criteria per the Data Management and Statistical core recommendations for the site
4. Must be willing to undergo all testing procedures, including neuroimaging and lumbar puncture.
5. Normal capacity to perform complex activities of daily living independently based on informant or physician report

Exclusion Criteria for Control Group

1. History of dream enactment behavior to suggest RBD
2. Parkinsonism, MSA, dementia, or mild cognitive impairment
3. Active central nervous system, systemic, psychiatric condition or use of psychoactive medication that would adversely affect cognitive, neuropsychiatric, motor, or autonomic functioning.
4. Contraindications to complete MRI.
5. Contraindications to lumbar puncture.
6. Participation in a clinical trial, except by specific permission by the Executive Committee
7. In the opinion of the investigator, the individual has a clinically significant uncontrolled medical condition that would impede safe completion of the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Idiopathic REM sleep behavior disorder, adults.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Prodromal Synucleinopathy Rating Scale | up to 5 years
  Rating scale combining neurocognitive battery, motor, autonomic, olfaction, color vision functions. Global score range 0-3, with higher score indicating greater symptoms of synucleinopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Yo-El Ju, MD, MCSI, Principal Investigator — Washington University School of Medicine; Brad Boeve, MD, Principal Investigator — Mayo Clinic; Ron Postuma, MD, Principal Investigator — McGill University
Locations (9):
- United States (8):
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Redwood City, California
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Oregon Health Sciences University, Portland, Oregon
- McGill University Health Centre Research Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified subject level data will be shared upon approved data request. This project will develop a large database of potential neurocognitive, neuroimaging, genetic, and polysomnographic biomarkers in rapid eye movement sleep behavior disorder (RBD), as well as a biobank of blood, DNA, RNA, and cerebrospinal fluid. A large part of the clinical battery is the Uniform Dataset version 3, will be uploaded to the National Alzheimer's Coordinating Center (NACC). Biofluid samples will be banked at the National Cell Repository for Alzheimer's Disease (NCRAD). Genetic data will be submitted to the National Institute on Aging Genetics of Alzheimer's Disease Data Storage (NIAGADS). Brain MRI and DaTscan imaging data will be uploaded to the Laboratory of NeuroImaging (LONI). Polysomnogram data will be uploaded to the National Sleep Research Resource (NSRR).
Supporting Information: Study Protocol
Time Frame: Updated datasets will be made available after completion of each semiannual data cleaning and data freeze. De-identified data will be available for at least the duration of the NAPS2 study.
Access Criteria: The NAPS2 Administrative Core will receive, process, and track all requests for data/biospecimens. All requests will be reviewed and tracked per the current NAPS Data Access Policy (https://www.naps-rbd.org/resources at the bottom of the webpage) at the time of request. Approved requests will be filled using data that has been de-identified.
URL: https://www.naps-rbd.org